CLINICAL TRIAL: NCT00404287
Title: Double Blind Randomized Phase IV Clinical Trial to Evaluate the Efficacy of Fluvastatin on Inflammatory Markers in the Haemodynamic Progression of Degenerative Aortic Stenosis. The AORTICA 1 Study.
Brief Title: Randomized Study to Evaluate the Efficacy of Fluvastatin on Inflammatory Markers in Patients With Aortic Stenosis.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not enough to complete the study
Sponsor: AORTICA Group (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, MD, PhD, AORTICA Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CXUO320BES04; EudraCT number 2005-003666-42
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Aortic Valve Stenosis
Keywords: C reactive protein; Inflammation; Aortic valve stenosis; progression
MeSH Terms: conditions — Aortic Valve Stenosis; Inflammation; Disease Progression | interventions — Fluvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fluvastatin (Active Comparator): fluvastatin 80 mg
  Interventions: Drug: Fluvastatin
- placebo (Placebo Comparator)
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
Atherosclerosis and aortic stenosis share inflammatory etiopathogenic characteristics in common. We hypothesized that statins therapy would decrease inflammatory markers concentrations in patients with degenerative aortic stenosis and halt the haemodynamic progression of the disease.

DETAILED DESCRIPTION:
This study will be a prospective, phase IV-III, randomized, double blinded, active controlled study, to evaluate the efficacy of fluvastatin on inflammatory markers in the haemodynamic progression of degenerative aortic stenosis. We hypothesized that statins therapy would decrease inflammatory markers concentrations in patients with degenerative aortic stenosis and halt the haemodynamic progression of the disease. Eligible patients with degenerative aortic stenosis will be randomized 1:1 to fluvastatin 80 mg once daily or placebo. The treatment should be continued until the study end (12 months). Follow up investigations will be performed after 3 months and at the end of the study (12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Asymptomatic
3. Aortic stenosis defined as aortic valve leaflet thickening with reduced systolic opening (maximum aortic jet velocity >2 m/s)
4. Written informed consent to participate in the study
5. Patients capable to follow all conditions along the study.

Exclusion Criteria:

1. Symptomatic patients caused by aortic stenosis.
2. Patients on statins anytime in the year before inclusion.
3. Patients diagnosed of dyslipidemia requiring statins.
4. Temperature ³37,8 ºC in the week before inclusion.
5. Any cardiovascular event succeeding in the three months before inclusion
6. Known thyrotoxicosis
7. Renal failure requiring hemodialysis
8. Any inflammatory noncardiac diseases or other reasons known to influence the study biomarkers concentrations.
9. Any surgery succeeding in the three months before inclusion.
10. Patients with any hepatopathy that in the view of the investigator prohibits participation in the study.
11. Patients with known muscular disease.
12. Patients with any severe medical condition that in the view of the investigator prohibits participation in the study
13. Use of corticoids, immunosuppressors or non steroid drugs.
14. Any known sensitivity to study drug (fluvastatin) or class of study drug.
15. Patients participating in any study in the last year.
16. Women of childbearing potential not using the contraception method(s) specified in this study, suspicion of pregnancy, as well as women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
To study changes in CRP (mg/dL) concentration at the end of the study (12 months) | 12 months

SECONDARY OUTCOMES:
To study changes in other inflammatory biomarkers (specify in the protocol) at the end of the study (12 months) | 12 months
To study changes in these biomarkers in the different grades of aortic stenosis at the end of the study (12 months) | 12 months
To study changes change in aortic valve area and medium aortic transvalvular gradient at the end of the study (12 months) | 12 months
To study the safety and tolerability of fluvastatin in patients with aortic stenosis. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Sanchez, MD, PhD, Principal Investigator — Hospital Universitario Gregorio Marañón de Madrid; Candido Martin-Luengo, MD, PhD, Study Chair — University of Salamanca
Locations (1):
- Hospital Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez PL, Mazzone A. C-reactive protein in degenerative aortic valve stenosis. Cardiovasc Ultrasound. 2006 Jun 14;4:24. doi: 10.1186/1476-7120-4-24. PMID 16774687
- [Background] Sanchez PL, Santos JL, Kaski JC, Cruz I, Arribas A, Villacorta E, Cascon M, Palacios IF, Martin-Luengo C; Grupo AORTICA (Grupo de Estudio de la Estenosis Aortica). Relation of circulating C-reactive protein to progression of aortic valve stenosis. Am J Cardiol. 2006 Jan 1;97(1):90-3. doi: 10.1016/j.amjcard.2005.07.113. Epub 2005 Nov 10. PMID 16377290